CLINICAL TRIAL: NCT07169162
Title: A Randomized, Double-blind, Parallel, Placebo-controlled, Flexible-dose Study of ADZENYS XR-ODT™ in Children Aged 4 to Less Than 6 Years Diagnosed With Attention-deficit/Hyperactivity Disorder (ADHD)
Brief Title: ADZENYS XR-ODT™ in Children (4 to <6 Years) Diagnosed With Attention-deficit/Hyperactivity Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment never started
Sponsor: Aytu BioPharma, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NT0202.1009
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine

STUDY DESIGN:
Intervention Model Description: Placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADZENYS XR-ODT (Experimental): Subjects will be assigned to receive ADZENYS XR-ODT orally disintegrating tablets in a randomized manner. Subjects will receive their dose once daily in the morning. All subjects will begin taking ADZENYS XR ODT 3.1 mg per day the morning after qualifying at Visit 2. The dose for each subject will be titrated in a stepwise fashion each week through Week 6 (Visit 8) based on the investigator's judgment of subject's clinical response (i.e., efficacy and tolerability) to 6.3 mg, 9.4 mg, 12.5 mg, 15.7 mg, up to 18.8 mg once daily, until an optimal dose or the highest dose is reached. No subject will receive a dose higher than 18.8 mg/day. Doses will comprise 1 or 2 tablets to achieve the (rounded) assigned dose. Once subjects reach an optimal dose of study drug, they will continue that dose for the remainder of the study.
  Interventions: Drug: ADZENYS XR-ODT
- Placebo (Placebo Comparator): Participants in this arm will be given placebo as matching ODT once daily during the double-blind treatment period.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: ADZENYS XR-ODT — ADZENYS XR-ODT™ (amphetamine) is an extended-release orally disintegrating tablet approved for once-daily oral administration for the treatment of ADHD in patients 6 years and older.
  Arms: ADZENYS XR-ODT
Drug: Placebo Oral Tablet — Participants in this arm will be given placebo as matching ODT once daily during the double-blind treatment period.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, flexible dose-titration, placebo-controlled, parallel-group study designed to evaluate the efficacy, safety, and tolerability of ADZENYS XR-ODT compared to placebo in children with ADHD.

DETAILED DESCRIPTION:
This randomized, double-blind, flexible-dose, placebo-controlled, parallel group study is designed to evaluate the efficacy, safety, and tolerability of ADZENYS XR-ODT compared to placebo in children with ADHD. Male and female children ages 4 to less than 6 years with a diagnosis of ADHD based on Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria (combined, inattentive, or hyperactive/impulsive) will be enrolled.

A Screening/Washout Period of up to 4 weeks (Days -28 to -1), which will include washout of any current ADHD medications (if applicable), will be followed by an 8-week, Randomized, Double-blind, Flexible-dose Period during which subjects will be randomly assigned to placebo or to ADZENYS XR-ODT once daily. All subjects will start on 3.1 mg of ADZENYS XR-ODT or matching placebo. The dose for each subject will be titrated in a stepwise fashion each week from Visit 3 to Visit 8 (Weeks 1 to 6) based on efficacy and tolerability to 6.3 mg; 9.4 mg; 12.5 mg; 15.7 mg; and 18.8 mg once daily, until an optimal dose or the highest dose is reached. No subject will receive a dose higher than 18.8 mg/day. Subjects must remain on a stable dose for at least 2 weeks.

An optimal dose is one that produces a reduction from Baseline of ADHD symptoms (ADHD Rating Scale IV [ADHD-RS-IV] Preschool Version) of ≥30% and a Clinical Global Impression Severity (CGI-S) score of 1 (normal), 2 (borderline ill), or 3 (mildly ill), while maintaining a tolerable adverse event (AE) profile. Once subjects reach an optimal dose of study drug, they will continue on that dose for the remainder of the study.

During titration, if a higher dose is not tolerated, the investigator may reduce the subject's dose by 1 dose level (this may not be done after Week 6 [Visit 8] of the study).

If further dose reductions are required, the subject should be discontinued from the study. Subjects who are unable to tolerate the lowest daily dose (3.1 mg) of study drug will be discontinued from the study.

Subjects who complete the 8-week Treatment Period may be eligible to enter the long-term safety and tolerability study of ADZENYS XR-ODT (NT0202.1010). For subjects to be eligible, they must complete Visit 10 without experiencing any clinically significant AEs that would preclude further exposure to ADZENYS XR-ODT. For subjects entering Study NT0202.1010, Visit 10 of this study can be Visit 1 of Study NT0202.1010, unless more than 2 weeks have elapsed since Visit 10. A safety follow-up telephone call will be made to parents/legal guardians approximately 1 week after discontinuation of study drug for subjects who do not roll over into Study NT0202.1010.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets DSM-5 criteria for ADHD, combined, hyperactive/impulsive, or inattentive presentation made during a clinical interview by an experienced clinician and confirmed with the K-SADS-PL.
* Subject has an age- and sex-adjusted rating of ≥90th percentile Total Score on the ADHD RS-IV Preschool Version (rated over past 6 months).
* Subject has a score of ≥4 on the CGI-S at Visit 2 (Baseline).
* Subject has had symptoms consistent with ADHD for at least 6 months.
* Subject has a Peabody Picture Vocabulary Test, 4th edition Standard Score of ≥70 at Visit 1 (Screening Visit).
* Subject has undergone an adequate course of nonpharmacological treatment for ADHD based on investigator judgment or the investigator considers the subject's condition severe enough to enroll without undergoing prior nonpharmacological treatment. Subjects who have been on a previous pharmacological treatment for ADHD may be enrolled provided they meet other entrance criteria.
* Subject has participated in structured group activity (e.g., preschool, daycare, camp) for at least 1 month that in the investigator's opinion allows assessment of symptoms and impairment in a setting outside of the home.

Exclusion Criteria:

* Other psychiatric diagnoses
* Significant cognitive impairment
* Chronic medical illnesses
* Structural cardiac defects
* Significant abnormal lab tests
* Taking disallowed medications
* Subject has history of or presence at Screening of long QT syndrome or QTc greater than 450 msec at Screening (using Fridericia's formula: QTcF) or any other clinically significant 12-lead ECG abnormality.
* Subject has a history of chronic vocal or motor tics or Tourette's syndrome or a family history of Tourette's syndrome.
* Subject has history or presence of suicidal ideation, significant self-injurious behavior, or violent behavior.
* Subject shows evidence of current physical, sexual, or emotional abuse.
* Subject has a height or a weight less than or equal to the 5th percentile for age and sex at the Screening Visit.
* Subject's blood pressure measurements exceed the 95th percentile for age, sex, and height at the Screening Visits (Visit 1) and/or Baseline Visit (Visit 2) per the American Academy of Pediatrics 2017 updated guidance.
* Subject's biological parent has a history of bipolar disorder.
* A parent/caregiver or someone living in the subject's home has a current or recent (past 12 months) history of substance abuse.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Attention-deficit/hyperactivity disorder Rating Scale-IV Preschool Version Total Score | Visit 10/Day 56
  Attention-Deficit/Hyperactivity Disorder Rating Scale-IV: Preschool Version (ADHD-RS-IV: Preschool Version) The ADHD-RS-IV Home and School checklists consist of the nine inattention and nine hyperactive/impulsive items that comprise the ADHD symptom criteria in the DSM-IV. Each item is rated on a four-point scale (0=never or rarely to 3=very often).
  Scores above the 93%ile are suspicious for but not diagnostic of preschool ADHD.
  Boys - Parent Inattention: 14 Hyperactivity/Impulsivity: 17 Total Score: 32/Teacher Inattention: 18 Hyperactivity/Impulsivity: 22 Total Score: 38 Girls - Parent Inattention: 12 Hyperactivity/Impulsivity: 14 Total Score: 24/Teacher Inattention: 11 Hyperactivity/Impulsivity: 13 Total Score: 24

SECONDARY OUTCOMES:
Clinical Global Impression - Severity | Visit 10/Day 56
Attention-deficit/hyperactivity disorder Rating Scale-IV Preschool Version Total Score | Visits 3-9 (Days 7, 14, 21, 28, 35, 42, 49)
Clinical Global Impression - Severity | Visits 3-9 (Days 7, 14, 21, 28, 35, 42, 49)

OTHER OUTCOMES:
Treatment-emergent adverse events, vital signs, clinical laboratory evaluations, and ECG results | Visits 3-9 (Days 7, 14, 21, 28, 35, 42, 49)
  Occurrence of treatment-emergent adverse events; specific evaluations of vital signs (oral or tympanic temperature, sitting blood pressure (taken in triplicate and averaged), pulse, and respiratory rate); height, weight, and body mass index clinical laboratory evaluations; and 12-lead electrocardiogram results
Children's Sleep Habits Questionnaire (CSHQ) Subscale and Total Sleep Disturbance Scores | Visits 3-9 (Days 7, 14, 21, 28, 35, 42, 49)
  The CSHQ is a psychological questionnaire designed to measure the most common sleep problems in children and adolescents 4 to 12 years of age. It contains items that relate to a number of key sleep domains that encompass the major sleep complaints in children and adolescents in this age group: bedtime behavior and sleep onset; sleep duration; anxiety around sleep; behavior occurring during sleep and night wakings; sleep-disordered breathing; parasomnias; and morning waking/daytime sleepiness.
  In the CSHQ, parents are asked to recall sleep behaviors that occur over a "typical" recent week. Items are rated on a 3-point scale: "usually" if the sleep behavior occurred 5 to 7 times per week; "sometimes" for 2 to 4 times per week; and "rarely" for 0 to 1 time/week.
  Although the entire CSHQ (Preschool and School-Aged) will be administered, the scoring will be done using the 33 Subscale items to provide Subscale and Total Sleep Disturbance scores.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn R Sikes, PhD, Study Director — Neos Therapeutics, Inc; Ann Childress, MD, Principal Investigator — Center for Psychiatry And Behavioral Medicine Inc.
Locations (1):
- Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided